CLINICAL TRIAL: NCT03765645
Title: Comparison of 9 Doses vs 3 Doses of Post Operative Antibiotics in Live Liver Donors: A Randomized Controlled Trial
Brief Title: Comparison of 9 Doses vs 3 Doses of Post Operative Antibiotics in Live Liver Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ILBS Liver Transplant 001
Record Dates: First submitted 2018-10-22; First posted 2018-12-05 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-02

CONDITIONS: Antibiotic Prophylaxis; Postoperative Infection
Keywords: Liver Transplant; Donor Hepatectomy; Antibiotic prophylaxis
MeSH Terms: interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3 doses on intra venous antibiotics (Active Comparator): Patients will receive 3 doses of intra venous antibiotics. (1 dose preoperative, 1 intra operative and 1 post-operative)
  Interventions: Drug: Piperacillin + Tazobactam
- 9 doses of intra venous antibiotics (Active Comparator): Patients will receive 9 doses of intra venous antibiotics. (1 dose preoperative, rest 8 doses at equal intervals)
  Interventions: Drug: Piperacillin + Tazobactam

INTERVENTIONS:
Drug: Piperacillin + Tazobactam — Antibiotic used will be Piperacillin + Tazobactam Dose: 4.5 g, thrice a day at regular intervals Route: Intra-venous

SUMMARY:
Antibiotic resistance is a very serious and dangerous situation in modern world. Judicious use of antibiotics is therefore of extreme importance not just in preventing antibiotic resistance but also it decreases cost of the treatment and prevent side-effects of the antibiotics. No randomized trial is available in literature for antibiotic prophylaxis in patient undergoing donor hepatectomy. Currently, antibiotic regimen is based on individual institutional protocol. There have been studies, comparing short course vs long dose of antibiotics in hepatectomy patients, concluding equivalent efficacy in preventing infective complications. The investigators aim at proving that 3 doses of antibiotics are equally effective in preventing infective complications, when compared to 9 doses of antibiotics, in patients undergoing donor hepatectomy. So, a randomized trial is required to study the antibiotic duration in patient undergoing donor hepatectomy.

DETAILED DESCRIPTION:
Antibiotic resistance is a very serious and dangerous situation in modern world. Judicious use of antibiotics is therefore of extreme importance not just in preventing antibiotic resistance but also it decreases cost of the treatment and prevent side-effects of the antibiotics. No randomized trial is available in literature for antibiotic prophylaxis in patient undergoing donor hepatectomy. Currently, antibiotic regimen is based on individual institutional protocol. So, a randomized trial is required to study the antibiotic duration in patient undergoing donor hepatectomy.

The investigators aim to prove that, in preventing infective complications, 3 doses of antibiotics are equally effective as compared to 9 doses of antibiotics in patients of donor hepatectomy.

Methodology:

The present study will be an equivalence randomized control trial where data will be collected from patients who are undergoing donor hepatectomy. Donor evaluation will be done according to institutional protocol. Donor evaluation will be done step wise as tabulated below.

Surgical technique After opening the abdomen through a J-shaped incision, cholecystectomy will be performed and intraoperative cholangiogram will be carried out through the cystic duct stump. The ipsilateral lobe will be mobilized and the hepatic vein will be looped. Hilar dissection will be performed and the ipsilateral portal vein and hepatic artery are defined. The transection plane will be determined by the line of demarcation obtained by temporary clamping of the ipsilateral portal vein and hepatic artery. Parenchymal transection will be performed without inflow occlusion by a Cavitron Ultrasonic Surgical Aspirator (CUSA_; Valleylab, Boulder, CO, USA). The last one-third of the transaction will be performed with a hanging maneuver. After completion of the transaction, the bile duct will be looped along with the sheath and a repeat cholangiogram will be performed by placing radio opaque markers at the proposed bile duct transection site. The bile duct will be divided between the markers. Intravenous heparin will be given (50 IU/kg); after waiting for 3 min, the hepatic artery, portal vein and hepatic vein will be divided between clamps and the graft will be taken out.

Assumptions:

* Prevalence of infective complications with 3 doses of antibiotic: 9%
* Prevalence of infective complications with 9 doses of antibiotic: 7% The alpha error, the power of the study and the equivalence margin will be taken as 5%, 80% and 15% respectively. For this investigators will need to enroll a total of 108 patients, equally divided into 2 groups.

Group A shall include 54 consecutive patients who are undergoing donor hepatectomy. These patients will be followed up closely in the post-operative period and would be serially sampled at pre-defined intervals. Patients will be assessed for infective complications. Antibiotics will be continued beyond 3 doses, if any sign of infection is present (Fever/ TLC more than 11,000/ Wound infection/others).

Group B shall include 54 patients, who will receive antibiotics for 3 days. These patients will also be followed up closely in the post-operative period and would be serially sampled at pre-defined intervals. Patients will be assessed for infective complications. Antibiotics will be continued beyond 3 days, if any sign of infection is present (Fever/ TLC more than 11,000/ Wound infection/others).

Infective complication rates / total duration of antibiotics/ cost of antibiotics and morbidity will be compared between the 2 cohorts.

EXPECTED OUTCOME: To establish that 3 doses of antibiotics are equally effective in preventing infective complications, as compared to 9 doses of antibiotics, in patients undergoing donor hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

• All patient undergoing donor hepatectomy consent for the study

Exclusion Criteria:

• Patients refusing consent for inclusion in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of infective complications | 1 year
  The number of infective complications (CDC guidelines) in post operative period will be compared among patients receiving 3 doses vs patients receiving 9 doses of antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Viniyendra Pamecha, Principal Investigator — ILBS
Locations (1):
- ILBS, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided